CLINICAL TRIAL: NCT01476319
Title: Improving Informed Consent Process for Percutaneous Cholecystostomy in the Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yen-Ko Lin, Attending Physician, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: KMUH-IRB-980360
Record Dates: First submitted 2011-08-01; First posted 2011-11-22 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis | interventions — Videotape Recording

ARMS (2):
- control (No Intervention)
- video (Experimental)
  Interventions: Other: video

INTERVENTIONS:
Other: video — The intervention group includes patients who obtain information about percutaneous cholecystostomy from a video will view at their bedside on a laptop.
  Arms: video

SUMMARY:
This study is planning to develop the audiovisual videos and determine whether educational videos are superior to routine discussion for informing patients in the emergency department (ED) about risks, benefits, and alternatives to receiving percutaneous cholecystostomy. Eligible patients will be approached when patients will be scheduled and waiting for receiving percutaneous cholecystostomy in the emergency department.

ELIGIBILITY:
Inclusion Criteria:

* All patients 18 years of age or older
* scheduled to receive the percutaneous cholecystostomy

Exclusion Criteria:

* clinically unstable
* refuse to participate
* are unable to understand the study process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-11-09 (Actual); Primary Completion 2014-09-09 (Actual); Study Completion 2014-09-09 (Actual)

PRIMARY OUTCOMES:
knowledge and satisfaction measure | immediately after intervention
  One questionnaire will be used as an outcome measure tool. Participants will be asked to complete one questionnaire with knowledge test and satisfaction evaluation with the process of informed consent after the educational sessions.

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung, Taiwan, Taiwan